CLINICAL TRIAL: NCT01734629
Title: Pulmonary Disease in Patients Referred for Coronary CT and Association Between Spirometric Abnormalities and Coronary Calcium Score.
Brief Title: Pulmonary Disease in Patients Referred for Coronary CT
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/02814-0 FAPESP; 0503/11 (Other: CAPPesq HCFMUSP)
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease; Atheroscleroses; COPD; Respiratory Diseases
Keywords: Coronary Disease; COPD; Spirometry; Coronary tomography
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Coronary CT Spirometry Cohort: Patients refereed to coronary CT enrolled in the study.

SUMMARY:
Several studies show an association between chronic obstructive pulmonary disease (COPD) and coronary artery disease (CAD). Besides risk factors such as smoking, both are associated with physical inactivity, advanced age and systemic inflammation The use of coronary computed tomography (CCT) with multiple detectors is a diagnostic method for coronary disease, describing the anatomy and severity of arterial obstruction. One way of estimating the cardiovascular risk is coronary calcium score (CCS). Due to the association between COPD and CAD, it is likely that many patients with IHD diagnosed by CT have reduced lung function.

The aim of this observational study is to establish the correlation between the CCS and lung function. It will also correlate the presence of irreversible airway obstruction with significant coronary lesions.

Patients over 40 years referred to CCT who agree to participate in the study will perform a spirometry with bronchodilator and collect a blood sample to measure serum markers of inflammation and cardiovascular risk (glycemia, lipid profile, C reactive protein (CRP), tumor necrosis factor-alpha (TNF-Alpha) and fibrinogen). The data will be compared in the general population and in subgroups: smokers, former smokers and nonsmokers.

One year after the CCT patients will be contacted by the investigators and accessed for emergency room visits, hospital admissions and fatal or nonfatal coronary or respiratory events.

The investigators hypothesis is that reduced lung function is independently associated with elevated CCS and is, also a risk factor for increased hospital admission and coronary events.

The concomitant assessment of lung function and CCS can contribute knowledge about the epidemiological association between pulmonary disease and CAD. This can also add to evidence for the use of spirometry as a marker of cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for coronary CT.
* Age greater than 40 years

Exclusion Criteria:

* History of myocardial revascularization (surgical or percutaneous)
* Cognitive-functional incapacity to perform spirometry
* Contraindication for administration of 400 mcg of albuterol
* Acute myocardial infarction or unstable angina within 2 weeks
* Angina pectoris class III or IV according to the Canadian Cardiovascular Society
* Heart failure New York Heart Association class III or IV

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 40 years old refereed to coronary CT in the investigator´s institution.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Coronary Calcium Score | Baseline
  Coronary calcium score is a measurement obtained in coronary computer tomography. The results will be compared between group with and without spirometric abnormalities.

SECONDARY OUTCOMES:
Coronary obstruction on CT | Baseline
  Presence or absence of coronary obstruction and it´s quantification by Duke score will be compared between group with and without spirometric abnormality.
Hospital Admissions | 1 year
  Hospital admissions will be accessed after one year from enrollment and compared between groups
ER visits | 1 year
  ER visits will be accessed after one year from enrollment and compared between groups
Fatal and non fatal cardiac or respiratory events | 1 year
  Fatal and non fatal cardiac or respiratory events will be accessed after one year from enrollment and compared between groups

OTHER OUTCOMES:
Smoking Status | 1 year
  All endpoints will be evaluated in smoking and nonsmoking subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Cukier, MD PHD, Principal Investigator — Incor - HCFMUSP
Locations (1):
- Heart Institute (InCor) do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Fernandes FLA, Carvalho-Pinto RM, Stelmach R, Salge JM, Rochitte CE, Souza ECDS, Pessi JD, Cukier A. Spirometry in patients screened for coronary artery disease: is it useful? J Bras Pneumol. 2018 Jul-Aug;44(4):299-306. doi: 10.1590/S1806-37562017000000276. PMID 30328928